CLINICAL TRIAL: NCT05361200
Title: Effects of Patient-Specific Adaptive Dynamic Cycling on Function Improvement in Individuals With Parkinson's Disease
Brief Title: Speed Manipulated Adaptive Rehabilitation Therapy Bike for Parkinson's Disease
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Responsible Party: Principal Investigator, Angela Ridgel, Professor, School of Health Sciences, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMARTPD
Record Dates: First submitted 2022-03-21; First posted 2022-05-04 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: movement disorders; exercise; adaptive therapy; cycling
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with 2 arms
Who Masked: Participant
Masking Description: Participant will not be told which group they were assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive dynamic cycling (Experimental): For the patient-specific adaptive dynamic cycling group, the optimization process will be done after the 3rd, 6th, and 9th sessions. The optimization procedure is based on sample entropy of cadence calculation from the previous session's cycling performance. After optimization, participants will receive specific settings for the next session.
  Interventions: Behavioral: Dynamic high-cadence cycling
- Non-adaptive dynamic cycling (Active Comparator): For the non-adaptive group, individuals will cycle on the dynamic bike with pre-determined settings that will stay constant throughout the exercise protocol.
  Interventions: Behavioral: Dynamic high-cadence cycling

INTERVENTIONS:
Behavioral: Dynamic high-cadence cycling — Resistance settings will be changed based on entropy of cadence every 3 sessions. Cadence will be set at 80RPM for both groups
  Other Names: S.M.A.R.T. cycling

SUMMARY:
Parkinson's disease (PD) is a progressive neurological disorder that results in slowness of movement, muscle stiffness, tremor, and postural instability. These symptoms significantly affect PD patients' quality of life, independence, and functional performance. There is currently no cure for PD, but symptoms can be treated with levodopa or deep brain stimulation surgery. Exercise-based rehabilitation has similar beneficial effects to surgical and pharmacological management without the potential negative side effects. Cycling-based interventions have been shown to increases motor function and mobility in individuals with PD. Specifically, benefits are greater when cycling cadence (revolutions per minute, RPM) is 30% greater than a self-selected pace.

Although high cadence cycling improves motor function in individuals with PD, there is significant heterogeneity in individual responses. To maximize the treatment effects and minimize the heterogeneity of high-cadence cycling, it is important to determine patient-specific settings. Previous studies have shown that higher variability (entropy) of cadence leads to greater improvement in motor function. The entropy of cadence calculation will be utilized to understand how patient-specific settings can drive improvements. The purpose of this study is to determine patient-specific settings and measure the effects of high cadence stationary (i.e. dynamic) cycling on functional performance in individuals with PD. Volunteers with Parkinson's disease will complete 12 cycling sessions over a 1-month period and measures of motor function, quality of life, functional performance, mood and exercise readiness will be collected.

DETAILED DESCRIPTION:
Potential participants will be prescreened with the ACSM pre-participation questionnaire over the phone or in person. Those who qualify will be asked to visit the research lab and sign the informed consent. Participants will be randomized into one of two groups: 1) patients-specific adaptive dynamic cycling or 2) non-adaptive dynamic cycling. Both groups will participate in a total of 12 sessions, each session consisting of 5 minutes of warm-up, 30 minutes of the main exercise, and 5 minutes of the cool-down period. For the patient-specific adaptive dynamic cycling group, the optimization process will be done after the 3rd, 6th, and 9th sessions. The optimization procedure is based on sample entropy of cadence calculation from the previous session's cycling performance. After optimization, participants will receive specific settings for the next session. For the non-adaptive group, individuals will cycle on the dynamic bike with pre-determined settings that will stay constant throughout the exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* 50-79 years of age
* no contraindications to exercise including cardiovascular disease or stroke

Exclusion Criteria:

* one or more major signs/symptoms of cardiovascular or pulmonary disease

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in motor symptoms | 4 weeks
  MDS-UPDRS Motor III (Movement Disorders Society- Unified Parkinson's Disease Rating Scale) Minimum Score-0 Maximum Score- 138 Lower score represents improvement
Change in motor kinematics | 4 weeks
  Kinesia One- Accelerometry- Lower score represents milder symptoms

SECONDARY OUTCOMES:
Change in quality of life | 4 weeks
  PDQ-39 (Parkinson' disease quality of life, 39 questions) Dimension score = sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100. Lower score reflect better QOL Minimum Score- 0 Maximum Score- 156
Change in mobility | 4 weeks
  Timed up and Go- Total time reported, lower time represents greater mobility

OTHER OUTCOMES:
Change in mood | 4 weeks
  Mood scales
Change in affect | 4 weeks
  Affective scales

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harper SA, Dowdell BT, Kim JH, Pollock BS, Ridgel AL. Non-Motor Symptoms after One Week of High Cadence Cycling in Parkinson's Disease. Int J Environ Res Public Health. 2019 Jun 14;16(12):2104. doi: 10.3390/ijerph16122104. PMID 31197095
- [Result] Mohammadi-Abdar H, Ridgel AL, Discenzo FM, Loparo KA. Design and Development of a Smart Exercise Bike for Motor Rehabilitation in Individuals with Parkinson's Disease. IEEE ASME Trans Mechatron. 2016 Jun;21(3):1650-1658. doi: 10.1109/TMECH.2015.2508030. Epub 2015 Dec 11. PMID 27298575
- [Result] Ridgel AL, Ault DL. High-Cadence Cycling Promotes Sustained Improvement in Bradykinesia, Rigidity, and Mobility in Individuals with Mild-Moderate Parkinson's Disease. Parkinsons Dis. 2019 Mar 3;2019:4076862. doi: 10.1155/2019/4076862. eCollection 2019. PMID 30944720
- [Result] Mohammadi-Abdar H, Ridgel AL, Discenzo FM, Phillips RS, Walter BL, Loparo KA. Test and Validation of a Smart Exercise Bike for Motor Rehabilitation in Individuals With Parkinson's Disease. IEEE Trans Neural Syst Rehabil Eng. 2016 Nov;24(11):1254-1264. doi: 10.1109/TNSRE.2016.2549030. Epub 2016 Mar 31. PMID 27046905